

May 17th, 2021

## **Statistical Analysis Plan and Preliminary Results**

**Hypothesis:** PE is predicted to be effective in reducing the EF and social impairments in these adolescents.

**Statistical Analysis:** Repeated measure ANOVA using SPSS ( is a software package used for interactive, or batched, statistical analysis) are performed to test the effectiveness of PE on social functions and EF in low and high autistic groups.

**Preliminary Results:** Reduced aggression for both autistic groups was found in the intervention when compared to control. Worse empathy in the intervention group when compared to the controls in both autistic groups.